CLINICAL TRIAL: NCT07255313
Title: Strengthening Psycho-physiological and Psycho-emotional Competencies in Healthcare Workers Through Mind Body Medicine and Nutrition: A Randomized Controlled Trial
Brief Title: Strengthening Health Literacy in Healthcare Workers Through Mind Body Medicine and Nutrition
Acronym: SOULFOOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Director of Research, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-12325-BO
Record Dates: First submitted 2025-11-17; First posted 2025-12-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Stress Resilience; Stress; Burnout; Burnout Syndrome
Keywords: stress resilience; work health promotion; burnout prevention; mental well-being; occupational stress; healthcare workers; Mind-Body Medicine; complementary medicine; nutrition; employee health; participatory research; randomized controlled trial; workplace intervention; self-care strategies; occupational health management; Self-Efficacy and Stress Resistance; nutrition and mental health
MeSH Terms: conditions — Burnout, Psychological; Psychological Well-Being; Occupational Stress

STUDY DESIGN:
Intervention Model Description: Intervention and control group with waitlist design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOULFOOD Programme (Experimental): This arm is a 10-week multimodal program designed to enhance resilience and health competencies. Participants engage in structured weekly intervention sessions lasting 2 hours and homework activities. These sessions are delivered in person, with flexible scheduling to accommodate work schedules. The intervention focuses on mind-body medicine, complementary medicine and nutrition. Core components include psycho-biotic nutrition, movement, relaxation techniques, and complementary self-care techniques. Each week covers a specific theme, such as mindful eating, emotional and stress regulation in the workplace, mindfulness, communication skills and social connections.
  Interventions: Behavioral: SOULFOOD Programme
- Waitlist Control Group (No Intervention): Participants in the waitlist control group do not receive any intervention during the 26-week waiting period. After this period, they will receive the same course program as the active intervention group.

INTERVENTIONS:
Behavioral: SOULFOOD Programme — This arm is a 10-week multimodal program designed to enhance resilience and health competencies. Participants engage in structured weekly intervention sessions lasting 2 hours and homework activities. These sessions are delivered in person, with flexible scheduling to accommodate work schedules. The intervention focuses on mind-body medicine, complementary medicine and nutrition. Core components include psycho-biotic nutrition, movement, relaxation techniques, and complementary self-care techniques. Each week covers a specific theme, such as mindful eating, emotional and stress regulation in the workplace, mindfulness, communication skills and social connections.
  Arms: SOULFOOD Programme

SUMMARY:
This is a randomized controlled trial aiming to develop and evaluate a workplace health program to improve stress resilience and mental well-being among healthcare workers at University Medicine Essen using a participatory research design (including a steering committee composed of hospital staff, needs assessment through focus groups, and pilot testing). The intervention combines mind-body medicine techniques, complementary medicine self-care strategies, and psycho-biotic nutrition. If successful, the program will be integrated into routine workplace health management and serve as a model for other healthcare institutions.

DETAILED DESCRIPTION:
This participatory research study at University Medicine Essen aims to develop, implement, and evaluate a workplace health program to improve stress resilience and mental well-being among healthcare workers. Increasing stress, staff shortages, and high rates of sick leave negatively impact both employees and patient care, making a comprehensive and sustainable health program essential. To ensure the intervention meets employees' needs, the study is guided by a steering committee consisting of hospital staff from various departments, including occupational health management, sustainability management, reintegration services, and the nonscientific staff council. A preliminary needs assessment will be conducted through focus groups, allowing employees to provide input on key aspects such as session format, duration, and content. Furthermore, the intervention design will be tested in a pilot phase to ensure the design is feasible and accepted by the participants.

The intervention will be a multimodal program combining mind-body medicine techniques, complementary self-care, and psycho-biotic nutrition to enhance stress resilience and overall health. Mind-body medicine includes mindfulness and stress management techniques, while complementary self-care will focus on easily applicable techniques from Traditional European Medicine (TEM) and Traditional Indian Medicine (TIM). Psycho-biotic nutrition, based on the connection between gut health and mental well-being, aims to support emotional and cognitive health through dietary changes. The study will use a randomized controlled trial design, comparing an intervention group with a waitlist control group to evaluate effectiveness.

Beyond individual benefits, the study also seeks to identify workplace-level improvements by promoting mindfulness among employees and leadership regarding structural stressors. This includes optimizing communication, understanding one's thoughts and emotions, and improving workplace policies such as break structures to better support employee well-being. By integrating feedback from the needs assessment and the pilot phase, the study aims to develop a sustainable and evidence-based health program that can be incorporated into routine workplace health management at University Medicine Essen. If successful, the intervention will serve as a model for other healthcare institutions and may be implemented more broadly within the healthcare sector.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Employees of University Medicine Essen
* Moderate resilience of ≤ 144 points on the RS-25
* Willingness to practice at home and keep a practice diary

Exclusion Criteria:

* Insufficient German language skills
* Pregnancy and breastfeeding
* Severe comorbid mental disorders (e.g., substance use disorder, major depression) or other severe comorbid somatic diseases (e.g., oncological disease without remission, severe pre-existing cardiovascular disease, organ failure, other severe neurological disorders)
* Planned or ongoing pension application (e.g., disability pension, occupational disability, reduced earning capacity, severe disability)
* Concurrent participation in other clinical intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Stress Resilience | Week 10
  Measured with the Resilience Scale (RS-25), a 25-item self-report instrument assessing personal competence and acceptance of life on one sum scale. Higher scores indicate greater resilience.

SECONDARY OUTCOMES:
Burnout | Week 10
  Assessed using the Maslach Burnout Inventory - Human Services Survey (MBI-HSS), a 22-item scale measuring emotional exhaustion, depersonalization, and personal accomplishment (three subscales). Higher exhaustion and depersonalization scores with lower personal accomplishment scores indicate a higher risk of burnout.
Stress Coping | Week 10
  Measured using the "Coping" subscale of the Stress- und Coping-Inventory (SCI-COPE), a 20-item self-report scale assessing five coping strategies on five subscales: positive thinking, active coping, social support, religion, and substance use (four items each). Higher scores indicate better coping skills.
Stress Symptoms | Week 10
  Measured using the "Symptoms"-subscale of the Stress- und Coping-Inventory (SCI-SYMPT), a 13-item self-report scale assessing physical and psychological stress symptoms (e.g., sleep disturbances, concentration issues). Higher scores indicate greater symptom burden on one sum scale.
Physical Resilience | Week 10
  Assessed with the subscale "Physical Resilience" of the Questionnaire for Assessing Health Behavior (FEG). It consists of five items rated on a Likert scale (1 = does not apply at all to 5 = fully applies), covering aspects such as perceived robustness, recovery after illness, and endurance in stressful situations. The mean of all items is calculated, with higher mean values indicating greater resilience.
Mental Well-Being | Week 10
  Measured with the World Health Organization (WHO-5) Well-Being Index, a self-report instrument measuring mental well-being. It consists of five statements summed up to one total scale. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being.
Psychological Distress | Week 10
  Psychological distress is assessed using the total score of the Patient Health Questionnaire-4 (PHQ-4), a brief self-report screening tool for anxiety and depressive symptoms. The PHQ-4 consists of four items rated on a 4-point Likert scale (0-3), yielding a total score ranging from 0 to 12. Higher scores indicate greater psychological distress.
Health Behaviour Change | Week 10
  This outcome measures participants' self-reported engagement in five domains of health-promoting behavior: relaxation, physical activity, breathing, nutrition, and complementary self-care. Assessment is conducted using the "Temple of Health," a pictorial tool consisting of five pillars representing these domains. Each pillar is 10 cm in height and serves as an visual analogue scale, with the bottom representing "I do not engage in this behavior" and the top representing "I fully engage in this behavior." Participants are instructed to color or draw on each pillar to indicate their perceived level of engagement.
Adverse Events | From enrollment to the end of treatment at week 10
  Adverse events are documented using participant self-report sheets provided at the beginning of the intervention period. Participants are instructed to record any physical or psychological complaints, discomfort, or other unexpected events that occur during the course of the study. Each entry includes the date, a brief description of the event, perceived severity, and whether the event is ongoing. The collected sheets are reviewed by the study team to identify, classify, and evaluate adverse events according to their frequency, severity, and potential relation to the intervention.
Stress Resilience | Week 26
  Measured with the Resilience Scale (RS-25), a 25-item self-report instrument assessing personal competence and acceptance of life on one sum scale. Higher scores indicate greater resilience.
Burnout | Week 26
  Assessed using the Maslach Burnout Inventory - Human Services Survey (MBI-HSS), a 22-item scale measuring emotional exhaustion, depersonalization, and personal accomplishment (three subscales). Higher exhaustion and depersonalization scores with lower personal accomplishment scores indicate a higher risk of burnout.
Stress Coping Strategies | Week 26
  Measured using the "Coping"-subscale of the Stress- und Coping-Inventory (SCI-COPE), a 20-item self-report scale assessing five different coping strategies on five subscales: positive thinking, active coping, social support, religion and substance use with four items each. Higher scores indicate better coping skills.
Stress Symptoms | Week 26
  Measured using the "Symptoms"-subscale of the Stress- und Coping-Inventory (SCI-SYMPT), a 13-item self-report scale assessing physical and psychological stress symptoms (e.g., sleep disturbances, concentration issues). Higher scores indicate greater symptom burden on one sum scale.
Physical Resilience | Week 26
  Assessed with the subscale "Physical Resilience" of the Questionnaire for Assessing Health Behavior (FEG). It consists of five items rated on a Likert scale (1 = does not apply at all to 5 = fully applies), covering aspects such as perceived robustness, recovery after illness, and endurance in stressful situations. The mean of all items is calculated, with higher mean values indicating greater resilience.
Mental Well-Being | Week 26
  Measured with the World Health Organization (WHO-5) Well-Being Index, a self-report instrument measuring mental well-being. It consists of five statements summed up to one total scale. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being.
Psychological distress | Week 26
  Psychological distress is assessed using the total score of the Patient Health Questionnaire-4 (PHQ-4), a brief self-report screening tool for anxiety and depressive symptoms. The PHQ-4 consists of four items rated on a 4-point Likert scale (0-3), yielding a total score ranging from 0 to 12. Higher scores indicate greater psychological distress.
Health Behaviour Change | Week 26
  This outcome measures participants' self-reported engagement in five domains of health-promoting behavior: relaxation, physical activity, breathing, nutrition, and complementary self-care. Assessment is conducted using the "Temple of Health," a pictorial tool consisting of five pillars representing these domains. Each pillar is 10 cm in height and serves as an visual analogue scale, with the bottom representing "I do not engage in this behavior" and the top representing "I fully engage in this behavior." Participants are instructed to color or draw on each pillar to indicate their perceived level of engagement.

OTHER OUTCOMES:
Mindfulness | Baseline
  Measured with the Mindful Attention Awareness Scale (MAAS), a 15-item self-report scale assessing everyday mindfulness. The mean of all items is calculated, with higher mean values indicating greater mindfulness in daily life.
Subjective Workload | Baseline
  Assessed using a Numeric Rating Scale (NRS), where participants rate their perceived workload on a scale from 0 (no burden) to 10 (maximum burden).
Ability to Change | Baseline
  The Perception, Intention and Ability to Change (PIAC) questionnaire is used to assess participants' perceived motivation and capability to initiate and implement health-related behavioral changes. It consists of nine items rated on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The items can be summarized to two subscales: perceptions and intentions regarding the need for change, and the perceived ability and implementation of behavioral changes. A total score is calculated by summing all items, with higher scores indicating a greater perceived internal ability to change.
Dietary Behavior | Baseline
  Assessed with the sum and subscores of the Eating Behavior (SEV) questionnaire, which assesses participants' self-reported eating behaviors and consists of two subscales: Health-Conscious Eating Behavior (GB-EV) and Weight-Controlled Eating Behavior (GK-EV). Items are rated on a 5-point Likert scale ranging from 1 (does not apply at all) to 5 (applies exactly). Higher scores indicate a stronger tendency toward health-conscious or weight-controlled eating behavior.
Physical Activity | Baseline
  Physical activity is assessed using the Movement and Sport Activity (BSA) questionnaire, which evaluates occupational, leisure-time, and sports-related activity on three subscales through a point-based scoring system. Occupational activity is calculated by combining sedentary, moderate, and vigorous activity items, with higher scores reflecting higher activity levels, resulting in an overall Occupational Physical Activity Index. Leisure-time activity is measured with frequency (days over the past four weeks) and duration (minutes per day) of eight activities to yield the Leisure-Time Physical Activity Index, Sport activity is assessed in the same manner, producing a Sports Activity Index in minutes per week. Higher index values indicate greater levels of physical activity.
Objective workload | Baseline
  Participants report the total number of hours they actually work per week. Data are collected via self-report. Higher values indicate a greater weekly workload.
Treatment expectations | Baseline
  This outcome assesses participants' expectations regarding how useful they believe the SOULFOOD program will be in strengthening their stress resilience. The measure is collected using a Numeric Rating Scale (NRS) ranging from 0 to 10, where 0 represents "not useful at all" and 10 represents "very useful". Higher scores indicate greater expectations.
Mindfulness | Week 10
  Measured with the Mindful Attention Awareness Scale (MAAS), a 15-item self-report scale assessing everyday mindfulness. The mean of all items is calculated, with higher mean values indicating greater mindfulness in daily life.
Subjective Workload | Week 10
  Assessed using a Numeric Rating Scale (NRS), where participants rate their perceived workload on a scale from 0 (no burden) to 10 (maximum burden).
Ability to Change | Week 10
  The Perception, Intention and Ability to Change (PIAC) questionnaire is used to assess participants' perceived motivation and capability to initiate and implement health-related behavioral changes. It consists of nine items rated on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The items can be summarized to two subscales: perceptions and intentions regarding the need for change, and the perceived ability and implementation of behavioral changes. A total score is calculated by summing all items, with higher scores indicating a greater perceived internal ability to change.
Dietary Behavior | Week 10
  Assessed with the sum and subscores of the Eating Behavior (SEV) questionnaire, which assesses participants' self-reported eating behaviors and consists of two subscales: Health-Conscious Eating Behavior (GB-EV) and Weight-Controlled Eating Behavior (GK-EV). Items are rated on a 5-point Likert scale ranging from 1 (does not apply at all) to 5 (applies exactly). Higher scores indicate a stronger tendency toward health-conscious or weight-controlled eating behavior.
Physical Activity | Week 10
  Physical activity is assessed using the Movement and Sport Activity (BSA) questionnaire, which evaluates occupational, leisure-time, and sports-related activity on three subscales through a point-based scoring system. Occupational activity is calculated by combining sedentary, moderate, and vigorous activity items, with higher scores reflecting higher activity levels, resulting in an overall Occupational Physical Activity Index. Leisure-time activity is measured with frequency (days over the past four weeks) and duration (minutes per day) of eight activities to yield the Leisure-Time Physical Activity Index, Sport activity is assessed in the same manner, producing a Sports Activity Index in minutes per week. Higher index values indicate greater levels of physical activity.
Objective workload | Week 10
  Participants report the total number of hours they actually work per week. Data are collected via self-report. Higher values indicate a greater weekly workload.
Mindfulness | Week 26
  Measured with the Mindful Attention Awareness Scale (MAAS), a 15-item self-report scale assessing everyday mindfulness. The mean of all items is calculated, with higher mean values indicating greater mindfulness in daily life.
Subjective Workload | Week 26
  Assessed using a Numeric Rating Scale (NRS), where participants rate their perceived workload on a scale from 0 (no burden) to 10 (maximum burden).
Ability to Change | Week 26
  The Perception, Intention and Ability to Change (PIAC) questionnaire is used to assess participants' perceived motivation and capability to initiate and implement health-related behavioral changes. It consists of nine items rated on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The items can be summarized to two subscales: perceptions and intentions regarding the need for change, and the perceived ability and implementation of behavioral changes. A total score is calculated by summing all items, with higher scores indicating a greater perceived internal ability to change.
Dietary Behavior | Week 26
  Assessed with the sum and subscores of the Eating Behavior (SEV) questionnaire, which assesses participants' self-reported eating behaviors and consists of two subscales: Health-Conscious Eating Behavior (GB-EV) and Weight-Controlled Eating Behavior (GK-EV). Items are rated on a 5-point Likert scale ranging from 1 (does not apply at all) to 5 (applies exactly). Higher scores indicate a stronger tendency toward health-conscious or weight-controlled eating behavior.
Physical Activity | Week 26
  Physical activity is assessed using the Movement and Sport Activity (BSA) questionnaire, which evaluates occupational, leisure-time, and sports-related activity on three subscales through a point-based scoring system. Occupational activity is calculated by combining sedentary, moderate, and vigorous activity items, with higher scores reflecting higher activity levels, resulting in an overall Occupational Physical Activity Index. Leisure-time activity is measured with frequency (days over the past four weeks) and duration (minutes per day) of eight activities to yield the Leisure-Time Physical Activity Index, Sport activity is assessed in the same manner, producing a Sports Activity Index in minutes per week. Higher index values indicate greater levels of physical activity.
Objective workload | week 26
  Participants report the total number of hours they actually work per week. Data are collected via self-report. Higher values indicate a greater weekly workload.
Adherence to Group Intervention | From enrollment to the end of treatment at week 10
  Adherence to the intervention program is assessed based on participants' attendance at each group session, marked as present or absent. Adherence is calculated as the proportion of attended sessions relative to the total number of scheduled sessions. Higher values indicate greater adherence to the course program.
Adherence to Home Work | From enrollment to the end of treatment at week 10
  Monitored through an adherence journal, where participants set personal goals related to mindful exercise, nutrition, relaxation, and complementary self-care strategies and earning points for daily use (as well as consistent engagement) outside of the group sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — University of Duisburg-Essen; Heidemarie Haller, PhD, Principal Investigator — University of Duisburg-Essen; Larissa Setzer, Principal Investigator — University of Duisburg-Essen
Locations (1):
- Center for Integrative Medicine and Planetary Health, University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographic information, baseline characteristics, outcome measures, and analyzable datasets used for primary and secondary endpoint analyses, will be made available to qualified researchers upon reasonable request and following review and approval by the study team.
Supporting Information: Study Protocol